CLINICAL TRIAL: NCT03573635
Title: Evaluation of the Effectiveness and Safety of an Own-invention System for Continuous Supraglottic Aspiration in Intubated and Mechanically Ventilated Patients: the "SUPRAtube" Device
Brief Title: Continuous Supraglottic Aspiration in Intubated and Mechanically Ventilated Patients: the "SUPRAtube" Device
Acronym: Supratube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 004
Record Dates: First submitted 2018-05-31; First posted 2018-06-29 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Aspiration Pneumonias
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supratube (Other): Patient with orotracheal intubation and supratube device
  Interventions: Device: Supratube; Other: Reference

INTERVENTIONS:
Device: Supratube — Aspiration of orotracheal secretions with supratube device
Other: Reference — Usual aspiration with any other device

SUMMARY:
Purpose of the trial: Evaluate the efficacy and safety of the device of self-invention of continuous oropharyngeal aspiration denominated "SUPRAtube" in patients with orotracheal intubation and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

• Endotracheal intubation and invasive mechanical ventilation,

Exclusion Criteria:

* Immediate postoperative oral cavity.
* Traumatic oral cavity injury.
* Platelet count less than 50000.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
aspirated secretions | 24 hours after intubation
  volume of aspirated secretions

SECONDARY OUTCOMES:
Adverse events | 24 hours after intubation
  Adverse events related to supratube device use

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Cardiovascular de Colombia, Piedecuesta, Santander Department, Colombia